CLINICAL TRIAL: NCT01805401
Title: Modulating Decision-Making and Impulse Control With Transcranial Direct Current Stimulation (tDCS) Over the Orbitofrontal Cortex (OFC): A Randomized and Sham-Controlled Study
Brief Title: tDCS Applied to the OFC: Effects on Decision-Making and Impulse Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Douglas Mental Health University Institute (Other)
Responsible Party: Principal Investigator, MARCELO T. BERLIM, Director, Neuromodulation Research Clinic, Douglas Mental Health University Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: REB-11/42; 2012 YIA (Other Grant/Funding Number: Brain & Behavior Research Foundation)
Record Dates: First submitted 2013-01-16; First posted 2013-03-06 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-10

CONDITIONS: Impulsive Behavior; Suicidal Impulses
Keywords: Decision-making; Impulse control; Transcranial direct current stimulation; Brain stimulation; Neuromodulation; tDCS; Iowa Gambling Task; Stroop Word-Color Task
MeSH Terms: conditions — Impulsive Behavior | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Left OFC Group (Experimental): Anode applied to the left OFC and cathode applied to the right OFC
  Interventions: Device: Transcranial Direct Current Stimulation
- Right OFC Group (Experimental): Anode applied to the right OFC and cathode applied to the left OFC
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham tDCS (Sham Comparator)
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Anode placed over the OFC or the DLPFC and cathode placed over the occipital region
  Other Names: tDCS, Brain Polarization

SUMMARY:
In this study the investigators aim to assess whether transcranial direct current stimulation (tDCS; a safe and non-invasive method for modulating the activity of specific brain regions) when applied over the orbitofrontal cortex (OFC) is able to modulate decision-making and impulse control in healthy participants.

DETAILED DESCRIPTION:
In this single-blind, three-arm and sham-controlled study, we will assess whether transcranial direct current stimulation (tDCS; a safe and non-invasive method for modulating the activity of specific brain regions) when applied over the orbitofrontal cortex (OFC) is able to modulate decision-making and impulse control in healthy volunteers. We hypothesize that tDCS applied to the OFC, in comparison to sham tDCS, will significantly enhance decision-making and impulse control. For this study we will enroll 45 healthy individuals aged 18-60 years. These individuals will be assessed with a battery of computerized tasks as well as clinician-administered and self-reported questionnaires on depression and anxiety. Assessments will be carried out before and after a single 30-minute tDCS session.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 to 60 years

Exclusion Criteria:

* Presence any psychiatric and/or neurological illness
* Psychoactive substance abuse/dependence in the past 6 months
* Current use of medication(s) that might influence cognition and/or affective status
* Presence of an uncontrolled medical disease (e.g., cardiovascular, renal)
* Pregnancy and/or lactation
* Specific contraindication for tDCS (e.g., metallic head implant).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2013-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in the net score of the Iowa Gambling Task | Before and after a 30-minute tDCS session

SECONDARY OUTCOMES:
Change in the "average-adjusted number of pumps" in the Balloon Analog Risk Task | Before and after a 30-minute tDCS session
Change in the number of risky choices in the Game of Dice Task | Before and after a 30-minute tDCS session
Change in the number of commission errors in the Continuous Performance Task | Before and after a 30-minute tDCS session
Change in the interference index in the Stroop Color-Word Test | Before and after a 30-minute tDCS session
Change in the stop-signal reaction time in the Stop-Signal Task | Before and after a 30-minute tDCS session

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Berlim, MD, MSc, Principal Investigator — Neuromodulation Research Clinic, Douglas Institute
Locations (1):
- Neuromodulation Research Clinic, Douglas Mental Health University Institute, Montreal, Quebec, Canada

REFERENCES:
- [Background] Beeli G, Casutt G, Baumgartner T, Jancke L. Modulating presence and impulsiveness by external stimulation of the brain. Behav Brain Funct. 2008 Aug 4;4:33. doi: 10.1186/1744-9081-4-33. PMID 18680573
- [Background] Boggio PS, Campanha C, Valasek CA, Fecteau S, Pascual-Leone A, Fregni F. Modulation of decision-making in a gambling task in older adults with transcranial direct current stimulation. Eur J Neurosci. 2010 Feb;31(3):593-7. doi: 10.1111/j.1460-9568.2010.07080.x. Epub 2010 Jan 25. PMID 20105234
- [Background] Fecteau S, Pascual-Leone A, Zald DH, Liguori P, Theoret H, Boggio PS, Fregni F. Activation of prefrontal cortex by transcranial direct current stimulation reduces appetite for risk during ambiguous decision making. J Neurosci. 2007 Jun 6;27(23):6212-8. doi: 10.1523/JNEUROSCI.0314-07.2007. PMID 17553993
- [Background] Hecht D, Walsh V, Lavidor M. Transcranial direct current stimulation facilitates decision making in a probabilistic guessing task. J Neurosci. 2010 Mar 24;30(12):4241-5. doi: 10.1523/JNEUROSCI.2924-09.2010. PMID 20335459
- [Background] Sela T, Kilim A, Lavidor M. Transcranial alternating current stimulation increases risk-taking behavior in the balloon analog risk task. Front Neurosci. 2012 Feb 14;6:22. doi: 10.3389/fnins.2012.00022. eCollection 2012. PMID 22347844